CLINICAL TRIAL: NCT02191189
Title: A Single-dose, 2-part, Open-label, Randomised, Pharmacoscintigraphic Investigation Into the Absorption of Nevirapine When Released Into Different Parts of the Gastro-intestinal Tract
Brief Title: Pharmacoscintigraphic Investigation Into the Absorption of Nevirapine When Released Into Different Parts of the Gastro-intestinal Tract in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1484
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (5):
- Treatment A, p.o. (Active Comparator): 50 mg Nevirapine administered orally in 100 mL water
  Interventions: Drug: Nevirapine suspension
- Treatment B, ascending colon (Experimental): 50 mg Nevirapine administered to the ascending colon via Enterion™ capsule
  Interventions: Drug: Nevirapine suspension, into Enterion™ capsule
- Treatment C, jejunum (Experimental): 50 mg Nevirapine administered to the jejunum via Enterion™ capsule
  Interventions: Drug: Nevirapine suspension, into Enterion™ capsule
- Treatment D, ileum (Experimental): 50 mg Nevirapine administered to the ileum via Enterion™ capsule
  Interventions: Drug: Nevirapine suspension, into Enterion™ capsule
- Treatment E, descending colon (Experimental): 50 mg Nevirapine administered to the descending colon via Enterion™ capsule
  Interventions: Drug: Nevirapine suspension, into Enterion™ capsule

INTERVENTIONS:
Drug: Nevirapine suspension, into Enterion™ capsule
  Arms: Treatment B, ascending colon; Treatment C, jejunum; Treatment D, ileum; Treatment E, descending colon
Drug: Nevirapine suspension
  Arms: Treatment A, p.o.

SUMMARY:
Study to determine the absorption of Nevirapine from different regions of the Gastro Intestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Aged 18-65 years
* Body Mass Index of between 18 and 35 kg/m2
* Subjects must be able to demonstrate ability to swallow an empty size 000 gelatin capsule
* Must be willing and able to participate in the whole study
* Must be able to provide signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months
* Those who are unable/unwilling to consume all the components of a standard meal or gelatine
* Subjects who have ever self referred or who have been referred to a physician or counsellor for abuse or misuse of alcohol, non-medical, medicinal drugs or other substance abuse e.g. solvents
* Any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD), and amphetamines (Class B unless prepared for injection, in which case amphetamines are Class A)
* Volunteers that admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months
* Positive drugs of abuse test result
* Regular alcohol consumption in males >= 21 units per week. (1 Unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine)
* Smoking of more than 10 cigarettes per day or equivalent (e.g. pipe, cigar, chewing tobacco)
* A breath carbon monoxide reading of greater than 20 ppm
* Inability to refrain from smoking for the duration of each study period
* Radiation exposure from clinical trials, including that from the present study and from diagnostic X-rays but excluding background radiation, exceeding 5 Millisieverts (mSv) in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Clinically significant abnormal biochemistry, haematology or urinalysis, as judged by the Investigator
* Liver function laboratory test (LFT) results outside the upper normal range. Subjects with LFTs > grade 1 will not be included
* History of gastrointestinal surgery, with the exception of appendicectomy unless it was performed within the previous 12 months
* History of clinically significant cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome
* History of chronic or acute infections
* Diseases of the central nervous system (such as epilepsy) and psychiatric or neurological disorders
* Acute diarrhoea or constipation in the 7 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion to be determined on first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
* Donation of blood within the previous three months
* Presence of non-removable metal objects such as metal plates, screws etc, in the abdominal region of the body
* Subjects will be excluded from the study if they are considered by the investigator to be at risk of transmitting through blood and other body fluids the agents responsible for AIDS (Acquired Immunodeficiency Syndrome) or other sexually transmitted disease or hepatitis. This will be achieved by the use of a card (similar to that used by the National Blood Transfusion Service), which asks a potential subject if they have reason to believe that they may fall into any category included on the card. If the verbal answer is in the affirmative then they will be excluded from the study.
* Positive hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV test results
* Subjects receiving prohibited medication. Subjects must not stop taking a prescribed medication for the purpose of entering the study.
* Failure to satisfy the Principal Medical Investigator of fitness to participate for any other reason

As a precaution, male subjects will be instructed to use appropriate barrier method contraception (e.g. condoms and spermicide) during the time interval between taking the first dose and three months following the last dose. Subjects will be advised to inform Pharmaceutical Profiles if their partner becomes pregnant within three months of them receiving the last dose of the study drug. Pharmaceutical Profiles will monitor the pregnancy to conclusion.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-05; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of nevirapine in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of nevirapine in plasma (Cmax) | up to 72 hours after drug administration
Time from dosing to the maximum concentration of nevirapine in plasma (tmax) | up to 72 hours after drug administration
Area under the concentration-time curve of nevirapine in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 72 hours after drug administration
Terminal elimination rate constant of nevirapine concentration in plasma (λz) | up to 72 hours after drug administration
Terminal half-life of nevirapine in plasma (t1/2) | up to 72 hours after drug administration
Mean residence time of nevirapine in the body after oral administration (MRTpo) | up to 72 hours after drug administration
Apparent clearance of nevirapine in the plasma after extravascular administration (CL/F) | up to 72 hours after drug administration
Apparent volume of distribution during the terminal elimination phase following an extravascular dose (Vz/F) | up to 72 hours after drug administration
Number of patients with adverse events | up to 78 days
Assessment of tolerability by investigator | Days 1-4 of each treatment period and at the end-of-study visit